CLINICAL TRIAL: NCT04885790
Title: Investigation of Dynamic Hyperinflation and Its Relationship With Functional Exercise Capacity in Children With Bronchiectasis
Status: Completed | Type: Observational
Sponsor: Izmir Bakircay University (Other)
Collaborators: Ege University (Other)
Responsible Party: Principal Investigator, Melih Zeren, Assist. Prof. Dr., Izmir Bakircay University
Other Study IDs: bakircaymzeren03
Record Dates: First submitted 2021-05-08; First posted 2021-05-13 (Actual); Last update posted 2021-10-25 (Actual); Status verified 2021-10

CONDITIONS: Bronchiectasis
Keywords: bronchiectasis; children; dynamic hyperinflation; exercise capacity; pulmonary function
MeSH Terms: conditions — Bronchiectasis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Bronchiectasis: Children with bronchiectasis
  Interventions: Other: Respiratory assessment using "Spiropalm 6MWT" portable spirometry; Other: Evaluation of functional exercise capacity; Other: Evaluation of peripheral muscle strength; Other: Evaluation of chronic cough

INTERVENTIONS:
Other: Respiratory assessment using "Spiropalm 6MWT" portable spirometry — "Spiropalm 6MWT" portable spirometry will be used during six-minute walk test for evaluation of dynamic hyperinflation and other related ventilatory parameters. The device will also be used as regular spirometry.
Other: Evaluation of functional exercise capacity — Functional exercise capacity of patients will be evaluated using six-minute walk test.
Other: Evaluation of peripheral muscle strength — Handgrip strength and M. Quadriceps strength will be evaluated using hand-held dynamometer.
Other: Evaluation of chronic cough — The Leicester Cough Questionnaire will be used for evaluating cough.

SUMMARY:
Prevalence of dynamic hyperinflation and its relationship with functional exercise capacity will be evaluated in children with bronchiectasis.

DETAILED DESCRIPTION:
Exercise or hyperpnea-induced air trapping is referred to as dynamic hyperinflation. In the presence of high resistance to expiratory flows and short expiratory times, the respiratory system is unable to return to its resting volume at the end of exhalation. The positive pressure within regions of hyperinflated lung raises the mean intrathoracic pressure and causes the inspiratory muscles to operate at a higher than resting lung volume. Thus, dynamic hyperinflation places the respiratory muscles at a considerable mechanical disadvantage and further impairs respiratory function. Dynamic hyperinflation is considered to be a key determinant of exercise capacity in patients with obstructive lung diseases. Although bronchiectasis is one of the obstructive lung diseases, the presence of dynamic hyperinflation in these patients has not been adequately investigated. Management guidelines of bronchiectasis state that imaging methods or pulmonary function tests alone is not sufficient to determine the disease burden and prognosis in these patients, so they recommend including detailed evaluation of exercise tolerance in the management of bronchiectasis. Aim of this study is to investigate the prevalence of dynamic hyperinflation and its relationship with functional exercise capacity in children with bronchiectasis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of bronchiectasis

Exclusion Criteria:

* Hospitalization history during past month
* Diagnosis of any other chronic childhood diseases such as cerebral palsy or neuromuscular diseases which may impede exercise tolerance

Ages: 8 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Children with bronchiectasis
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-08-10 (Actual); Study Completion 2021-08-10 (Actual)

PRIMARY OUTCOMES:
Dynamic hyperinflation | At baseline
  Dynamic hyperinflation will be defined as a decrease of >100 mL in inspiratory capacity at the end of six-minute walk test determined by Spiropalm 6MWT device.

SECONDARY OUTCOMES:
Six-minute walk distance | At baseline
  Distance walked in six minutes will be recorded. Test will be conducted according to the guideline of American Thoracic Society.
Minute ventilation | At baseline
  Maximum minute ventilation during six-minute walk test will be measured via Spiropalm 6MWT device.
Breathing reserve | At baseline
  Breathing reserve (BR) will be calculated as the difference between the maximal voluntary ventilation (MVV) and the maximum minute ventilation (VE) as a fraction of the MVV using Spiropalm 6MWT during six-minute walk test.
Forced Vital Capacity (FVC) | At baseline
  FVC will be measured before six-minute walk test according to the guideline of European Respiratory Society.
Forced Expiratory Volume in 1 second (FEV1) | At baseline
  FEV1 will be measured before six-minute walk test according to the guideline of European Respiratory Society.
Peak Expiratory Flow (PEF) | At baseline
  PEF will be measured before six-minute walk test according to the guideline of European Respiratory Society.
Handgrip strength | At baseline
  Handgrip strength will be measured using handgrip dynamometer.
M. Quadriceps strength | At baseline
  M. Quadriceps strength will be measured using hand-held dynamometer
Leicester Cough Questionnaire | At baseline
  Chronic cough will be evaluated using Leicester Cough Questionnaire. Questionnaire consists of 19 items covering physical, psychological and social domains with a 7 point likert response scale (range from 1 to 7). Higher score indicates better quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Ege University Faculty of Medicine, Department of Pediatrics, Division of Pediatric Pulmonology, Izmir, Turkey (Türkiye)